CLINICAL TRIAL: NCT05562843
Title: Autologous Cellular Therapy With PRP-PC in Chronic Lung Diseases: An Observational Study LI-004
Acronym: PRP-PC
Status: Completed | Type: Observational
Sponsor: H-CYTE (Industry)
Responsible Party: Sponsor
Other Study IDs: HCYTE LI-004
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: COPD ILD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Autologous Cellular Therapy with PRP-PC — In this study, cells will be harvested from the patient from the peripheral blood, isolated and concentrated using centrifugation, then returned to the patient same day via the peripheral circulation.

SUMMARY:
For this study, cells will be harvested from the patient from the peripheral blood, isolated and concentrated using proprietary Emcyte™ equipment/centrifugation, and then returned to the patient same day via the peripheral circulation. As circulation occurs, the concentrated cells enter the right heart and are then disseminated into the lungs, becoming trapped in the lung's microcirculation. Here, the cells are believed to produce multiple bioactive factors such as cytokines and anti-inflammatory mediators. Several growth factors are released by activated platelets becoming honing cells for healing within the tissue. The exact long-term mechanism of action of PRP-PC in the lungs remains under investigation. Safety studies have proven that autologous treatment is incredibly safe, largely because of the minimal cell manipulation and the autologous nature of the cells. Prior observational studies in this are have shown strong safety profiles as well as strong efficacy in both COPD and ILD.

DETAILED DESCRIPTION:
Study Objective(s) Primary

* To determine if pulmonary function improves following ceullar therapy Secondary
* To determine if participants' perceived quality of life related to breathing improves following cellular therapy To evaluate the safety of autologous PRP-PC administration for chronic lung disease

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 and older
2. Diagnosis of COPD or an interstitial lung disease

Exclusion Criteria:

Pregnant subjects, subjects with an active cancer diagnosis except for basal cell skin cancer-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Conventional treatment for chronic lung disease typically involves inhaled bronchodilators, steroids, oxygen therapy, antifibrotic medications, lung reduction surgery and lung transplantation for the management of symptoms, although none of these modalities (aside from surgery/transplant) thwarts long-term progression of the disease.. With transplantation the availability of donor lungs is scarce and the longterm need for anti-rejection medication and monitoring can be overwhelming. Recent advances in the field of regenerative medicine in lung disease have demonstrated that autologous cellular therapy may reduce inflammation and aid in the maintenance and repair of damaged lung tissue
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary Lung Function | 3 months
  Lung function will be measured with spirometry to test FVC volume, FVC % predicted, FEV1 volume, and FEV1% predicted.

SECONDARY OUTCOMES:
Quality of Life subjective | 3 and 12 months
  Quality of life will be measured with the Clinical COPD Questionnaire (CCQ).

CONTACTS AND LOCATIONS:
Locations (1):
- Centers for Respiratory Health, Tampa, Florida, United States